CLINICAL TRIAL: NCT06606522
Title: A Diagnostic System of Clincial Model and Urinary Biomarkers for Intrinsic Acute Kidney Disease
Brief Title: A Clinical Diagnostic System for Intrinsic Acute Kidney Disease
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Affiliated Hospital of Hebei University (Other); Beijing Miyun Hospital (Unknown); Dongzhimen Hospital, Beijing (Other); Taiyuan Central Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, Peking University First Hospital
Other Study IDs: 2024-379-002
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Disease
Keywords: acute kidney disease; kidney biopsy; diagnostic model; urinary biomarkers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine samples from patients with acute kidney disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Derivation cohort: Patients from Peking University First Hospital
  Interventions: Diagnostic Test: Clinical model; Diagnostic Test: Urinary biomarkers
- External Validation Cohort: Patients from other four centers
  Interventions: Diagnostic Test: Clinical model; Diagnostic Test: Urinary biomarkers

INTERVENTIONS:
Diagnostic Test: Clinical model — Clinical model: a clinical model based on basic demorgraphic information and commonly executed laboratory tests to differentiate different pathological types of intrinsic AKD.
Diagnostic Test: Urinary biomarkers — Urinary biomarkers: biomarkers help differentiate different pathological types of intrinsic AKD.

SUMMARY:
The goal of this observational cross-sectional study is to develop a clinical diagnostic system for intrinsic acute kidney disease (AKD) to help clincians make non-invasive diagnosis when a kidney biopsy is not available. The main questions it aims to answer are:

1. Can a clinical model comprised of common clinical indexes help diagnose AKD ?
2. Can a combinition of several urinary biomarkers help diagnose AKD ? The study will be conducted in retrospective cohorts of patients with AKD undergoing kidney biopsy. The gold standard of the study is histological diagnosis of AKD. The model will be developed in a derivation cohort from one center, and will be further externally validated in a multicent cohort. The urinary biomarkers will only be tested in the derivation cohort.

DETAILED DESCRIPTION:
Acute kidney disease is a frequent syndrome characterized by a sudden loss of kidney function. AKD caused by intrinsic kidney diseases are usually more severe than other causes. The treatment of intrinsic AKD mostly depends on a definite pathological diagnosis, requiring invasive kidney biopsy which is not available in all AKD cases. The goal of this study is to develop a clinical diagnostic system comprised of clinical model and urinary biomarkers for intrinsic AKD to help clincians make non-invasive diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with AKD undergoing kidney biopsy between Jan. 1, 2020 and Dec. 31, 2024.

Exclusion Criteria:

* Patients were excluede if they

  1. underwent a biopsy to evaluate renal allograft rejection;
  2. had a history of hematopoietic stem cell transplantation;
  3. were diagnosed with hematological malignancy or end-stage tumor with kidney metastasis;
  4. were tested antineutrophil cytoplasmic autoantibody (ANCA) or double-strand DNA (dsDNA) or anti-glomerular basement membrane (GBM) antibody positive before biopsy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with AKD undergoing kidney biopsy between Jan. 1, 2020 and Apr. 30, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1360 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Histological diagnosis of AKD | within a week after biopsy
  Number of definite biopsy-proven histological diagnosis of AKD

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, Professor, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Dongzhimen Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Miyun District Hospital, Beijing, Beijing Municipality
  - Affliated Hospital of Hebei University, Baoding, Hebei
  - Taiyuan Central Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No